CLINICAL TRIAL: NCT07277998
Title: Clinical Efficacy of Alternating Intralesional Triamcinolone Acetonide and Platelet-Rich Plasma Compared to Triamcinolone Alone in Patients With Oral Submucous Fibrosis: A Two-Arm Interventional Clinical Trial
Brief Title: Alternating Triamcinolone and Platelet-Rich Plasma Therapy for Oral Submucous Fibrosis
Acronym: RegenOSF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karachi Medical and Dental College (Other)
Responsible Party: Principal Investigator, Madiha Khan, Principal Investigator, Karachi Medical and Dental College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MK_OSF_ALTTA_PRP_2025; KMDC/OMFS/OSF-CombTherapy/2025 (Other: Karachi Medical and Dental College)
Record Dates: First submitted 2025-11-27; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Oral Submucous Fibrosis
Keywords: Triamcinolone acetonide; Platelet-rich plasma; Regenerative therapy; Oral mucosal disorders; Fibrosis; OSF; Intralesional therapy; Oral and maxillofacial surgery; Steroid injection; Mouth opening; Burning sensation; Oral precancerous lesions; Stem cell mediated healing; Collagen remodeling; Areca nut; Trismus; Limited mouth opening; LMO; BMS; OMFS; Regenerative dentistry; Oral surgery; PRP
MeSH Terms: conditions — Oral Submucous Fibrosis; Fibrosis; Paresthesia; Trismus | interventions — Injections; Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: Two-arm parallel assignment comparing alternating-week Triamcinolone + PRP therapy vs standard single-agent therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alternating Triamcinolone + PRP Therapy (Active Comparator): Patients will receive alternating-week intralesional Triamcinolone (10 mg/mL) and Platelet-Rich Plasma therapy. Triamcinolone is given in Week 1, PRP in Week 2, and alternated weekly for a total of 6-8 sessions.
  Interventions: Biological: Platelet-Rich Plasma (PRP) Injections; Drug: Triamcinolone Acetonide
- Triamcinolone Alone Therapy (Active Comparator): Patients will receive intralesional Triamcinolone acetonide (10 mg/mL) once weekly for 6-8 sessions as standard therapy.
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Biological: Platelet-Rich Plasma (PRP) Injections — Autologous Platelet-rich plasma (PRP) injected intralesionally at standard volume for Oral submucous fibrosis (OSF) treatment, administered every alternate week.
  Other Names: PRP
  Arms: Alternating Triamcinolone + PRP Therapy
Drug: Triamcinolone Acetonide — Triamcinolone acetonide 10 mg/mL administered intralesionally once weekly.
  Other Names: TA

SUMMARY:
Oral Submucous Fibrosis (OSF) is a chronic, progressive, potentially malignant disorder characterized by mucosal stiffness, trismus, and burning sensation. This interventional clinical trial evaluates the therapeutic effectiveness of alternating weekly intralesional Triamcinolone Acetonide (TA) and Platelet-Rich Plasma (PRP) injections compared to standard Triamcinolone therapy alone. The purpose is to determine whether sequential anti-inflammatory (TA) and regenerative (PRP) stimulation can produce superior clinical improvement in mouth opening, burning sensation, and mucosal flexibility compared to corticosteroid therapy alone.

DETAILED DESCRIPTION:
Oral Submucous Fibrosis (OSF) is a chronic, irreversible fibro-elastic disorder of the oral mucosa associated with restricted mouth opening, burning sensation, impaired mastication, and decreased quality of life. Traditional management approaches include intralesional corticosteroids, physiotherapy, antioxidants, and more recently, regenerative therapies such as Platelet-Rich Plasma (PRP).

Triamcinolone Acetonide (TA) provides anti-inflammatory and anti-fibrotic effects by suppressing fibroblast activity and collagen deposition. PRP, an autologous concentrate of platelets and growth factors, has demonstrated potential in promoting angiogenesis, collagen remodeling, and mucosal regeneration. Alternating TA and PRP may theoretically combine the immediate anti-inflammatory benefits of TA with the long-term regenerative benefits of PRP, resulting in more effective improvement of OSF symptoms.

This study consists of two arms. In the control arm, participants will receive weekly intralesional Triamcinolone injections for 6 weeks. In the experimental arm, participants will receive Triamcinolone in Week 1, PRP in Week 2, followed by alternating TA and PRP injections for a total of 6 weeks. All participants will be instructed to perform standardized jaw physiotherapy exercises during the study period.

Primary outcomes include change in interincisal mouth opening (millimeters) and reduction in burning sensation using a Visual Analog Scale (VAS). Secondary outcomes include mucosal flexibility score, cheek rigidity grading, functional improvement during mastication and speech, and patient satisfaction.

This clinical trial aims to generate high-quality comparative evidence regarding whether an alternating TA-PRP protocol offers superior therapeutic outcomes compared to conventional corticosteroid therapy alone, thereby supporting advancement of regenerative treatment protocols for OSF within oral and maxillofacial clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Clinically diagnosed Oral Submucous Fibrosis (OSF), Stage II-IV using Haider et al. classification.

Age 18-65 years. Mouth opening ≤ 30 mm. Persistent burning sensation (VAS ≥ 3). Able and willing to comply with weekly therapy sessions. Provided written informed consent.

Exclusion Criteria:

Previous treatment with PRP, Platelet-rich Fibrin (PRF), corticosteroid, or combination therapy in the last 6 months.

Systemic diseases affecting wound healing (e.g., uncontrolled diabetes, severe anemia).

Current steroid therapy or immunosuppressive therapy.

Oral lesions suspicious for malignancy or recurrent Oral Squamous cell carcinoma (OSCC).

Bleeding disorders or platelet count <150,000.

Pregnant or breastfeeding women.

Known allergy to local anesthetics or triamcinolone.

Patients unwilling to stop areca nut/tobacco habits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Mouth Opening (Interincisal Distance in mm) | Baseline, Week 4, Week 8, Week 12
  Mouth opening will be measured using a digital caliper from incisal edge to incisal edge at baseline and at each follow-up visit. The primary endpoint is the change in interincisal distance from baseline to 8 weeks and 12 weeks.
Change in Burning Sensation (VAS Score 0-10) | Baseline, Week 4, Week 8, Week 12
  Burning sensation will be assessed using the Visual Analog Scale (VAS), where 0 indicates no burning and 10 indicates the worst possible burning.

SECONDARY OUTCOMES:
Change in Clinical Grade of OSMF | Baseline and Week 12
  Oral Submucous Fibrosis (OSF) severity will be assessed using a standardized clinical grading system that evaluates mouth opening, fibrous banding, mucosal texture, and burning sensation. Grades range from Grade I (mild) to Grade IV (severe). Higher grades indicate more advanced disease. Improvement or worsening will be determined by comparing baseline and Week 12 assessment
Change in Cheek Flexibility (mm) | Baseline, Week 8, Week 12
  Cheek flexibility will be measured using Mathur and Jha method at baseline and follow-up visits.
Incidence of Treatment-Related Adverse Events | Up to 12 weeks
  All adverse events such as swelling, pain, ulceration, infection, or allergy will be recorded throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Sufyan Ahmed, BDS, FCPS, Study Chair — Karachi Medical and Dental College
Locations (1):
- Abbasi Shaheed Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset will be used for future analyses, internal audits, and subsequent publications by the study team. Data will remain confidential and securely stored according to institutional policy.

REFERENCES:
- [Result] Khan M, Ahmed S, Faraz A, Ali Z, Khan S, Iqbal M. Comparison Between Treatment of Oral Submucous Fibrosis with Intralesional Triamcinolone Injection Versus Platelet-Rich Plasma. Journal of Population Therapeutics and Clinical Pharmacology. 2025;32(4):166-172.
- [Result] Alsousou J, Thompson M, Hulley P, Noble A, Willett K. The biology of Platelet-Rich Plasma and regenerative potential in tissue healing. Am J Sports Med. 2009;37(11):2259-2272. PMID: 19088268.
- [Result] Tilakaratne WM, Klinikowski MF. Intralesional corticosteroid injection as a treatment modality for oral submucous fibrosis. J Oral Pathol Med. 2016;45(3):162-168. PMID: 27422421.
- [Result] Saraf K, Gaur A, Thomas R. Efficacy of Platelet-Rich Plasma injections in Oral Submucous Fibrosis: A Prospective Clinical Study. Dent Res Dent Clin Dent Prospects. 2021;15(4):275-280. PMID: 34912641.
- [Result] OSF Singh S, Misra N. Comparative evaluation of intralesional platelet-rich plasma and intralesional corticosteroid in management of oral submucous fibrosis. J Oral Maxillofac Pathol. 2020;24(1):121-126. PMID: 33584414.
- [Result] Ali H, Ahmed S, Raza SH. Effect of intralesional injection of triamcinolone acetonide in oral submucous fibrosis. Journal of Surgery Pakistan. 2019;24(4):181-185.
- [Result] Haider SM, Merchant A, Fida M. Clinical grading of oral submucous fibrosis: A practical classification for patient severity assessment. Journal of Pakistan Dental Association. 2016;25(4):147-152.
- See also: Published comparative study on PRP and TA therapy for Oral Submucous Fibrosis by the Principal Investigator. — https://www.jptcp.com/index.php/jptcp/article/view/10065
- See also: Institutionally developed OSF clinical grading system used in this trial. — https://pubmed.ncbi.nlm.nih.gov/10783440/
- See also: Steroid-based management study of Oral Submucous Fibrosis conducted at the same institution. — https://www.jsp.org.pk/index.php/jsp/article/view/170?utm_source=chatgpt.com